CLINICAL TRIAL: NCT02412969
Title: Impact of Dural Puncture Epidural Versus Traditional Lumbar Epidural on Onset of Labor Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Latha Hebbar, Professor and Director of OB Anesthesia, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00034219
Record Dates: First submitted 2014-08-22; First posted 2015-04-09 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Labor Pain; Labor Analgesia
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lumbar Epidural (Active Comparator): Control group will have standard of care Lumbar Epidural
  Interventions: Procedure: Lumbar Epidural
- Dural Puncture Epidural (Experimental): Will receive Dural Puncture Epidural
  Interventions: Procedure: Dural Puncture Epidural

INTERVENTIONS:
Procedure: Lumbar Epidural — control group will receive lumbar puncture epidural
  Arms: Lumbar Epidural
Procedure: Dural Puncture Epidural — intervention group will receive a dural puncture epidural
  Arms: Dural Puncture Epidural

SUMMARY:
This study is to examine the onset of pain relief with two different methods of labor epidural. The traditional labor epidural involves the placement of numbing and anti-pain medicine in the epidural space which surrounds the spinal cord. In order to take effect, the medication has to cross a layer of tissue called the dura. In the current study, the same medications are placed in the epidural space after the dura is punctured with a fine needle. This research, will help evaluate whether this technique will result in earlier onset of pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients in active painful labor
* ASA I and II parturients
* Women Ages 18+ to 40
* Patients who have labor epidural as part of their labor plan will be recruited

Exclusion Criteria:

* Patients admitted to the Labor and Delivery Suite who are committed to have a delivery with the current admission but who do not want a labor epidural
* Patients with the following: bleeding disorders, infection at the site of epidural placement, generalized sepsis, stenotic heart valve lesions, increased intracranial pressure, patients with hypovolemia, and patient refusal
* Parturients with chronic pain syndromes
* Patients on MAO inhibitors
* Patients with allergies to bupivacaine and fentanyl (and other amide local anesthetics) patients with substance abuse history will be excluded
* Non English-speaking patients will be excluded

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2014-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Compare time of onset of labor analgesia Dural Puncture vs Lumbar Puncture | two days post delivery

SECONDARY OUTCOMES:
Incidence of Side Effect | two days post delivery
  Incidence of maternal motor block, hypotension, pruritis, headache, patient satisfaction and fetal bradycardia.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States